CLINICAL TRIAL: NCT01889914
Title: Treatment by Subcutaneous Continuous Infusion of Insulin by Portable Pump Versus Discontinuous Infusion of Insulin by Multi-injections in the Type 2 Diabetes: Study of the Insulinosensibility in the 2 Types of Treatments
Brief Title: TReatment by Insulin Continuous Infusion in Type 2 DIAbetes
Acronym: TRICIDIA2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-004602-19
Record Dates: First submitted 2013-06-06; First posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous infusion of insulin by pump (Experimental): in this arm called "continuous infusion of insulin with a pump" the patient receive continuous rapid insulin (APIDRA ®)with an external pump.
  An hepatic IRM and a botnia test will be practice before and six months after the beginning of this treatment(continuous insulin)
  Interventions: Drug: 2 different procedures of administration of insulin
- discontinuous insulin multiple injections (Experimental): An arm called " intensification of the multiple daily injections ": the patient will receive an additional injection of basal insulin LEVEMIR® : five injections per day (2 injections of Levemir® and 3 injections of Apidra®) instead of four previously (1 injection of Levemir® and 3 injections of Apidra®).
  An hepatic IRM and a botnia test will be practice before and six months after the beginning of the treatment
  Interventions: Drug: 2 different procedures of administration of insulin

INTERVENTIONS:
Drug: 2 different procedures of administration of insulin — Compare the efficiency of both types of therapeutic care in insulinoresistant type 2 diabetic patients: insulin multi injections (levemir et Apidra versus continuous infusion of insulin apidra by pump
  Other Names: multiple daily discontinuous injections of insulin; continuous infusion of rapid insulin by an external pump

SUMMARY:
The aim of the TRICIDIA2 study is to compare two modalities of administration of insulin.

In our future study, the investigators wish to study if the treatment by continuous infusion of insulin improves the insulinosensitivity of type 2 diabetic patients; the investigators indeed expect that the insulin delivered in a continuous way decreases the insulino-resistance of these patients compared with the intermittent delivering of insulin.

DETAILED DESCRIPTION:
We wish to use before and after treatment the classic tools of measure of insulinosensitivity / the euglycemic hyperinsulinemic clamp associated with a measure of the insulinosecretion thanks to a test of load in glucose IV. The coupling in the same procedure of these 2 tests is the Botnia clamp. We also wish to use the continuous measure of subcutaneous glucose during several days to estimate the reduction in the average glycemia on the fast and prandial periods as well as the decrease of the time spent in hyperglycemia during the day. This tool demonstrated its interest in type 2 diabetic population in several studies. Finally the current / spectro-IRM methods of imaging are now validated to quantify and measure exactly the importance of the steatosis, including in type 2 patients, because we know that it is probably the result of the insulino-resistance; We would also like to demonstrate that some genetic polymorphisms of proteins (polymorphisms G / T493 of the MTP, 1927 C/T of the receiver R1 of the adiponectin and 265 C/T of the gene of Apolipoprotéines A) are factors which can modulate the steatosis development in case of type 2 diabetes.

In other secondary criteria we wait for an improvement of HbA1c, quality of life of type 2 obese people with regard to the treatment by intensified Multi-injections.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* type 2 diabete patient with insuline basal/bolus treatment for at least 6 months
* Doses of insuline > 0,7 U/Kg/j
* HbA1c ≥ 7,5%
* without ADO for at least 4 weeks (sulfamides, Incrétines, glinides, acarbose) except the metformine
* BMI ≥ 28,5 kg/m²
* clinical diagnostique of diabetes for at least 10 ans
* Patient must be able to Realize an automonitoring and to manage the functioning of an insulin pump.

Exclusion Criteria:

* glitazone treatment less than 3 month before inclusion
* Patient with an untreated by the laser proliferative ischemic retinopathy
* BMI < 28,5 kg/m²
* Pacemaker (CI IRM)
* Presence of implantable material (CI IRM)
* Pregnancy, breast-feeding
* Practices of violent sports
* Professional extreme environment of cold or heat
* Serious psychiatric diseases physical and/or psychiatric Incapacitated medically significant
* Poor sanitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-03 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
changes from baseline in insulinoresistance measured by biological tests of hyperinsulinemic euglycemic clamp in the two groups of treatment 6 months after the start of the treatment. | baseline and six months after the begining of the study

SECONDARY OUTCOMES:
change from baseline in the hyperglycemia time spent during basal and prandial period with continuous glucose monitoring tool at 6 months | baseline and six months after the beginning of the study
change from baseline in HbA1c in the two groups of treatment at three, six, nine and twelve months | baseline and three, six, nine, twelve months
change from baseline in quality of life measured with questionnaires at 6 months | baseline and 6 months
change from baseline in weight at three, six, nine and twelve months in the two groups. | baseline and three, six, nine and twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Sabine RUDONI, MD, Principal Investigator — CHU de BOCAGE, DIJON, FRANCE
Locations (1):
- CHU, Dijon, France